CLINICAL TRIAL: NCT01814878
Title: A Randomized, Active-Controlled, Parallel Group, Double-Blind Study to Compare the Efficacy and Safety of Tramadol HCl/Acetaminophen ER and IR in Subjects Who Complain of Moderate to Severe Postoperative Pain
Brief Title: A Study Comparing the Effectiveness and Safety of Extended Release (ER) Tramadol Hydrochloride (HCl)/Acetaminophen With Immediate Release (IR) Tramadol HCl/Acetaminophen in Participants With Moderate to Severe Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR016636; TRAMAPPAI3005
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Tramadol Hydrochloride; Acetaminophen; Ultracet
MeSH Terms: conditions — Pain, Postoperative | interventions — Ultracet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol Hydrochloride/Acetaminophen ER (Experimental): Participants will be administered 2 oral tablets of extended release (ER) tramadol HCl (75 milligram [mg])/acetaminophen (650 mg) and 2 tablets of placebo matching to immediate release (IR) tramadol HCl/acetaminophen orally every 12 hours up to 36 hours, and 2 tablets of placebo matching to IR tramadol HCl/acetaminophen every 6 hours up to 42 hours.
  Interventions: Drug: Tramadol HCl/Acetaminophen ER
- Tramadol HCl/Acetaminophen IR (Active Comparator): Participants will be administered 2 oral tablets of IR tramadol HCl (37.5 mg)/acetaminophen (325 mg) and 2 tablets of placebo matching to ER tramadol HCl/acetaminophen at 0, 12, 24 and 36 hours, and 2 tablets of IR tramadol HCl/acetaminophen at 6, 18, 30 and 42 hours.
  Interventions: Drug: Tramadol HCl/Acetaminophen IR

INTERVENTIONS:
Drug: Tramadol HCl/Acetaminophen ER — 2 tablets of ER (tramadol HCl [75 mg]/acetaminophen [650 mg]) will be administered at 0, 12, 24 and 36 hours
  Other Names: Ultracet
  Arms: Tramadol Hydrochloride/Acetaminophen ER
Drug: Tramadol HCl/Acetaminophen IR — 2 tablets of IR (tramadol HCl [37.5 mg]/acetaminophen [325 mg]) at 0, 6, 12, 18, 24, 30, 36 and 42 hours
  Other Names: Ultracet
  Arms: Tramadol HCl/Acetaminophen IR

SUMMARY:
The purpose of this study is to compare the efficacy and safety of extended release (ER) tramadol hydrochloride (HCl)/acetaminophen with immediate release (IR) tramadol HCl/acetaminophen in participants with moderate to severe (very serious, life threatening) postoperative pain.

DETAILED DESCRIPTION:
This study is a randomized (study drug assigned by chance), multicenter (when more than 1 hospital or medical school team work on a medical research study), active-controlled, parallel group (each group of participants will be treated at the same time), double-blind (neither physician nor participant knows the treatment that the participant receives) study. The duration of the treatment will be 2 days and will be conducted in 4 periods: screening period (from 33 to 2 days before study drug administration to the first surgical incision), surgical period (to 1 day before study drug administration), qualification period (1 day) and double-blind treatment period (1 to 2 days). Participants will be randomly assigned to 2 groups: study drug treatment group (ER) and comparator treatment group (IR). Participants will be administered 2 tablets of ER tramadol HCl (75 milligram [mg])/acetaminophen (650 mg) along with 2 tablets of placebo matching to IR tramadol HCl/acetaminophen in study drug treatment group; and 2 tablets of IR tramadol HCl (37.5 mg)/acetaminophen (325 mg) along with 2 tablets of placebo matching to ER tramadol HCl/acetaminophen in comparator treatment group respectively at 0, 12, 24 and 36 hours. Participants will also be administered 2 tablets of placebo matching to IR tramadol HCl/acetaminophen in study drug treatment group; and 2 tablets of IR tramadol HCl/acetaminophen in comparator treatment group respectively at 6, 18, 30 and 42 hours. Participants will be administered investigational product at 6-hour interval from the time of the first investigational product administration over 48 hours. Efficacy will be assessed using 11-point numeric rating scale (NRS). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are scheduled to have standard primary (non-revision) unilateral (having to do with only 1 side of a structure) total knee replacement arthroplasty (TKRA-surgery to fix a joint) for non-inflammatory (no swelling, redness, and pain in tissues caused by injury or damage) degenerative joint disease (NIDJD)
* Participants who are capable of oral (having to do with the mouth) intake
* Women must be: postmenopausal (for at least 1 year), surgically sterile, abstinent (not having sexual intercourse), or practicing a highly effective method of birth control before participation in the study and who agree to continue to use the same method of birth control throughout the study in cases of women of childbearing potential
* Male participants must practice contraception, and must agree not to donate his sperms for 1 month after the last dose of study drug
* Participants who will complain of baseline pain of intensity of greater than or equal to 4 on 11-point numeric rating scale (NRS) measured within 1 hour prior to randomization (study drug assigned by chance) and a maximum of 6 hours after discontinuation of participant controlled analgesia (PCA) after at least 12 hours of application following TKRA

Exclusion Criteria:

* Participants with Illness history (severe [very serious, life threatening] hepatic [having to do with the liver] failure, severe renal [having to do with the kidney] failure; severe respiratory depression; risk for mental fog with head injury or brain lesions [abnormal area of tissue, such as a wound, sore, rash, or boil]; digestive ulcer [sore], severe blood abnormalities; severe cardiac insufficiency; aspirin asthma [asthmatic attack-breathing disorder in which there is a wheezing and difficulty in breathing; caused by non-steroidal anti-inflammatory drugs] or history of aspirin asthma; history of epilepsy [seizure disorder]; rheumatism, significant psychiatric disorder or taking antipsychotic drugs for psychiatric treatment)
* Administration of disallowed therapy such as: administration of oral, patch, injection or local analgesics (drug used to control pain) acting centrally (the brain and the spinal cord) or peripherally (not central) before study drug administration after completion of PCA application, surgery is conducted simultaneously in addition to TKRA, administration of monoamine oxidase (MAO) inhibitors or discontinuation of the administration within 2 weeks, tricyclic antidepressants that may increase the seizure (sudden, uncontrolled muscle spasms and loss of consciousness resulting from abnormal brain function) risk when concomitantly (given at the same time) administered, neuroleptics, or drugs that may lower the seizure threshold, use of sedatives (a medication to calm or make less anxious) other than that used for general anesthesia (loss of sensation or feeling) during surgery
* Participants who used any study drug or investigational medical device within 30 days before the start of the treatment
* Participants requiring postoperative intensive care unit (ICU) care
* Participants having hypersensitivity to tramadol or acetaminophen

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea Ltd. Clinical Trial, Study Director — Janssen Korea Ltd.

REFERENCES:
- [Derived] Park YB, Ha CW, Cho SD, Lee MC, Lee JH, Seo SS, Kang SB, Kyung HS, Choi CH, Chang N, Rhim HY, Bin SI. A randomized study to compare the efficacy and safety of extended-release and immediate-release tramadol HCl/acetaminophen in patients with acute pain following total knee replacement. Curr Med Res Opin. 2015 Jan;31(1):75-84. doi: 10.1185/03007995.2014.975338. Epub 2014 Oct 31. PMID 25299350

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride (HCl)/Acetaminophen ER: Participants received 2 oral tablets of extended-release (ER) tramadol HCl (75 milligram [mg])/acetaminophen (650 mg) and 2 tablets of placebo matched to immediate-release (IR) tramadol HCl/acetaminophen orally every 12 hours up to 36 hours, and 2 tablets of placebo matched to IR tramadol HCl/acetaminophen every 6 hours up to 42 hours.
- Tramadol HCl/Acetaminophen IR: Participants received 2 oral tablets of IR tramadol HCl (37.5 mg)/acetaminophen (325 mg) and 2 tablets of placebo matched to ER tramadol HCl/acetaminophen at 0, 12, 24 and 36 hours, and 2 tablets of IR tramadol HCl/acetaminophen at 6, 18, 30 and 42 hours.
Period: Overall Study
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Started | 162 | 158
Completed | 116 | 128
Not Completed | 46 | 30
Not completed — Adverse Event | 16 | 5
Not completed — Withdrawal by Subject | 20 | 16
Not completed — Protocol Violation | 5 | 5
Not completed — Physician Decision | 3 | 1
Not completed — Screening failure (drop-out) | 0 | 3
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR | Total
Number analyzed (Participants) | 162 | 158 | 320
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (6.4) | 67.5 (6.6) | 67.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 138 | 293
  Male | 7 | 20 | 27

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference (SPID) at Hour 48
Description: The SPID is time-weighted sum of all observations of pain intensity difference (PID) collected at each measurement time point from Baseline to 48 hours. PID: Baseline pain intensity (PI) minus current PI; PI was assessed using 11-point numeric rating scale (NRS, 0=no pain to 10=worst pain imaginable). PI score ranges from 0-3 where 0=no pain and 3=severe pain. PI score of 0=NRS score of 0, PI score of 1=NRS score >=1 and <=3, PI score of 2=NRS score of >=4 and <=6 and PI score of 3=NRS score of >=7 and <=10. Total score for SPID at 48 hours (SPID48) ranges from -144 (worst) to 144 (best).
Time Frame: Hour 48
Population: The per-protocol (PP) population included all randomly assigned participants who did not violate major eligibility criteria and whose SPID was calculated with actual measurements or adjusted values at all assessment time points.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 139 | 127
Units on scale | 32.5 (30.7) | 37.2 (23.9)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Non-inferiority comparison for Tramadol Hydrochloride/Acetaminophen ER to Tramadol HCl/Acetaminophen IR was performed; Test type: Non-Inferiority or Equivalence — Study drug treatment group was considered non-inferior to comparator treatment group, if lower limit of the confidence interval was larger than -2.0; p = 0.1648, Student's t-test — Hour 48: P-value was calculated using Student's t-test; Mean Difference (Final Values) = -4.68, 95% CI 2-sided [-11.29 to 1.93]

2. Secondary Outcome: Sum of Pain Intensity Difference (SPID) at Hour 6, 12 and 24
Description: The SPID is time-weighted sum of all observations of PID collected at each measurement time point from Baseline to 24 hours. PID: Baseline PI minus current PI; PI was assessed using 11-point NRS, 0=no pain to 10=worst pain imaginable. PI score ranges from 0-3 where 0=no pain and 3=severe pain. PI score of 0=NRS score of 0, PI score of 1=NRS score >=1 and <=3, PI score of 2=NRS score of >=4 and <=6 and PI score of 3=NRS score of >=7 and <=10. Total score ranges from -18 (worst) to 18 (best) for SPID6, -36 (worst) to 36 (best) for SPID12 and -72 (worst) to 72 (best) for SPID24.
Time Frame: Hour 6, 12, 24
Population: The intent-to-treat population included all randomly assigned participants. Here, 'N' (number of participants analyzed) specifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 162 | 155
Units on scale
  Hour 6 | 3.6 (3.7) | 3.9 (3.3)
  Hour 12 | 7.0 (7.8) | 8.1 (6.5)
  Hour 24 | 14.6 (15.3) | 17.6 (12.7)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.4082, Student's t-test — Hour 6: P-value was calculated using Student's t-test; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-1.10 to 0.45]
Statistical Analysis 2: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1720, Student's t-test — Hour 12: P-value was calculated using Student's t-test; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-2.68 to 0.48]
Statistical Analysis 3: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.0589, Student's t-test — Hour 24: P-value was calculated using Student's t-test; Mean Difference (Final Values) = -2.99, 95% CI 2-sided [-6.09 to 0.11]

3. Secondary Outcome: Total Pain Relief (TOTPAR) Score
Description: Pain relief was measured on a 5-point categorical scale of 0-4 (0=no change, 1=slight relief, 2=moderate relief, 3=fair relief, 4=pain resolved completely). TOTPAR was calculated as the time-weighted sum over all pain relief up to 48 hours. Total score ranges from 0 (worst) to 24 (best) for TOTPAR6, 0 (worst) to 48 (best) for TOTPAR12, 0 (worst) to 96 (best) for TOTPAR24 and 0 (worst) to 192 (best) for TOTPAR48.
Time Frame: Hour 6, 12, 24, 48
Population: The intent-to-treat population included all randomly assigned participants. Here, 'N' specifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 161 | 151
Units on scale
  Hour 6 | 6.0 (4.8) | 6.8 (5.7)
  Hour 12 | 12.5 (10.4) | 14.7 (11.1)
  Hour 24 | 27.1 (21.3) | 31.0 (22.5)
  Hour 48 | 55.6 (43.2) | 61.7 (44.5)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1542, Student's t-test — Hour 6: P-value was calculated using Student's t-test
Statistical Analysis 2: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.0714, Student's t-test — Hour 12: P-value was calculated using Student's t-test
Statistical Analysis 3: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1147, Student's t-test — Hour 24: P-value was calculated using Student's t-test
Statistical Analysis 4: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.2209, Student's t-test — Hour 48: P-value was calculated using Student's t-test

4. Secondary Outcome: Sum of Total Pain Relief and Sum of Pain Intensity Difference (SPRID)
Description: The SPRID is sum of SPID and TOTPAR. In SPID, PI score ranges from 0-3 where 0=no pain and 3=severe pain. PI score of 0=NRS score of 0, PI score of 1=NRS score >=1 and <= 3, PI score of 2=NRS score of >=4 and <=6 and PI score of 3=NRS score of >=7 and <=10. In TOTPAR, pain relief score ranges from 0-4 (0=no change, 1=slight relief, 2=moderate relief, 3=fair relief, 4=pain resolved completely). Total score ranges from -18 (worst) to 42 (best) for SPRID6, -36 (worst) to 84 (best) for SPRID12, -72 (worst) to 168 (best) for SPRID24 and -144 (worst) to 336 (best) for SPRID48.
Time Frame: Hour 6, 12, 24, 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 161 | 151
Units on scale
  Hour 6 | 9.6 (7.3) | 10.9 (8.1)
  Hour 12 | 19.6 (15.7) | 23.1 (15.2)
  Hour 24 | 41.8 (31.6) | 49.1 (30.8)
  Hour 48 | 85.9 (64.7) | 97.0 (61.0)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1498, Student's t-test — Hour 6: P-value was calculated using Student's t-test
Statistical Analysis 2: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.0485, Student's t-test — Hour 12: P-value was calculated using Student's t-test
Statistical Analysis 3: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.0404, Student's t-test — Hour 24: P-value was calculated using Student's t-test
Statistical Analysis 4: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1210, Student's t-test — Hour 48: P-value was calculated using Student's t-test

5. Secondary Outcome: Time to the First Rescue Medication Administered Because of Insufficient Pain Relief
Description: The time until administration of the first rescue medication (rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation) because of insufficient pain relief after administration of the study drug was recorded. Rescue medications allowed were oral or injection of tramadol HCl (intramuscular [directly into muscle] or intravenous injection [directly into vein]).
Time Frame: Baseline up to Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 29 | 30
Minutes | 1339 (710) | 1212 (853)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.4216, Wilcoxon (Mann-Whitney) — P-value was calculated using Mann-Whitney's U test

6. Secondary Outcome: Number of Doses of Rescue Medication Administered Because of Insufficient Pain Relief
Description: The frequency of the rescue medication (rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation) because of insufficient pain relief was measured after administration of the study drug. Rescue medications allowed were oral or injection of tramadol HCl (intramuscular or intravenous injection).
Time Frame: Baseline up to Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 29 | 30
Doses | 2.1 (1.9) | 1.4 (0.9)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.1000, Wilcoxon (Mann-Whitney) — P-value was calculated using Mann-Whitney's U test

7. Secondary Outcome: Dosage of Rescue Medication Administered Because of Insufficient Pain Relief
Description: The dosage of the rescue medication (rescue medications are medicines that are administered to the participants when the efficacy of the study drug is not satisfactory, or the effect of the study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation) because of insufficient pain relief was measured after administration of the study drug. Rescue medications allowed were oral or injection of tramadol HCl (intramuscular or intravenous injection).
Time Frame: Baseline up to Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Milligram
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 29 | 30
Milligram | 50.0 (0.0) | 51.7 (9.1)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.3255, Wilcoxon (Mann-Whitney) — P-value was calculated using Mann-Whitney's U test

8. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: The PGIC was used to assess the degree of participant's overall improvement with treatment, and participants were instructed to assess how much the overall status had been improved after investigational product administration compared to baseline in 7 grades (1=Very much improved and B=Very much worsened).
Time Frame: Day 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Number analyzed (Participants) | 134 | 138
Units on scale | 2.71 (0.86) | 2.60 (0.80)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride (HCl)/Acetaminophen ER vs Tramadol HCl/Acetaminophen IR; Test type: Superiority or Other; p = 0.2848, Student's t-test — Day 3: P-value was calculated using student's t-test

ADVERSE EVENTS:
Time Frame: Screening up to Day 3 or early withdrawal
Description: Safety population included all participants who received at least 1 dose of study drug. Number of participants evaluable for safety was 161 in Tramadol Hydrochloride/Acetaminophen ER arm and 153 in Tramadol HCl/Acetaminophen IR arm.
Arm/Group | Tramadol Hydrochloride (HCl)/Acetaminophen ER | Tramadol HCl/Acetaminophen IR
Serious Adverse Events (participants affected / at risk) | 1/161 | 0/153
Other Adverse Events (participants affected / at risk) | 139/161 | 129/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride (HCl)/Acetaminophen ER (N=161) | Tramadol HCl/Acetaminophen IR (N=153)
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride (HCl)/Acetaminophen ER (N=161) | Tramadol HCl/Acetaminophen IR (N=153)
Constipation (Gastrointestinal disorders) | 39 | 30
Dyspepsia (Gastrointestinal disorders) | 11 | 20
Nausea (Gastrointestinal disorders) | 80 | 68
Vomiting (Gastrointestinal disorders) | 45 | 37
Pyrexia (General disorders) | 28 | 36
Wound secretion (Injury, poisoning and procedural complications) | 11 | 6
Haemoglobin decreased (Investigations) | 38 | 40
Dizziness (Nervous system disorders) | 17 | 13
Headache (Nervous system disorders) | 15 | 9
Dysuria (Renal and urinary disorders) | 27 | 24
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 26
Somnolence (Nervous system disorders) | 9 | 8
Insomnia (Psychiatric disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is cancelled.